CLINICAL TRIAL: NCT07081737
Title: The Future of Pain Management: Can Person-centred and Precision AI-Based Decision Support Enhance Interdisciplinary Rehabilitation for Chronic Pain?
Brief Title: Person-Centred AI Support in Interdisciplinary Rehabilitation for Chronic Pain
Acronym: pAIn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bjorn Ang (Other)
Collaborators: Göteborg University (Other); Forte (Industry); Dalarna County Council, Sweden (Other); Karolinska Institutet (Other); The Swedish Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Bjorn Ang, Professor, Dalarna University
Organization: Dalarna University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-04532-01
Record Dates: First submitted 2024-01-23; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Pain, Chronic; Chronic Pain, Widespread; Pain Management
Keywords: chronic pain; prediction; Artificial Intelligence; Interdisciplinary pain rehabilitation; Machine learning; Clinical Decision Support System (CDSS)
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: A two-armed, multi-site cluster randomized controlled trial (2026-2029) will be conducted across 20 interdisciplinary rehabilitation clinics. Clinics are randomized to standard interdisciplinary treatment (IDT) with or without a Clinical Decision Support System (CDSS). The design follows the UK Medical Research Council (MRC) framework for complex interventions and includes a pilot RCT, a full-scale effectiveness and cost-utility trial, and a concurrent process evaluation. Patients are recruited via routine care. Outcomes are assessed at baseline, post-IDT, and 12-month follow-up. Primary outcome: a patient-prioritized composite of health-related well-being. Secondary outcomes: SF-36, EQ-5D, HADS, WAI, and register-based data on sickness absence and medication (followed for 5 years). Cost-utility (QALYs, ICERs) and implementation (using Normalization Process Theory) are evaluated.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary treatment (IDT) + Clinical Decision Support System (CDSS) (Experimental): Participants in this arm receive standard interdisciplinary treatment (IDT) for complex chronic pain, supported by a Clinical Decision Support System (CDSS). The CDSS provides individualized prognostic and predictive outputs using advanced AI-clustered models trained on linked national registry data. Clinicians access the CDSS through a secure interface integrated into clinical workflows, offering data-driven support for person-centred treatment planning and goal setting. The intervention is designed to enhance decision-making, treatment precision, and long-term outcomes such as work ability, well-being, and quality of life. The CDSS is used by the care team prior to and during the rehabilitation program.
  Interventions: Other: Interdisciplinary treatment (IDT) + Clinical Decision Support System (CDSS)
- Interdisciplinary treatment (IDT) (Active Comparator): Participants in this control-arm receive standard interdisciplinary treatment (IDT) for complex chronic pain. IDT is delivered by a coordinated team of healthcare professionals-typically including physicians, psychologists, physiotherapists, and occupational therapists-and is based on evidence-informed rehabilitation protocols. The program emphasizes biopsychosocial assessment, goal setting, and individually tailored interventions aimed at improving function, coping, and quality of life. No use of the Clinical Decision Support System (CDSS) is included in this arm.
  Interventions: Other: Interdisciplinary treatment (IDT)

INTERVENTIONS:
Other: Interdisciplinary treatment (IDT) + Clinical Decision Support System (CDSS) — Interdisciplinary treatment (IDT) combined with Clinical Decision Support System (CDSS)
  Arms: Interdisciplinary treatment (IDT) + Clinical Decision Support System (CDSS)
Other: Interdisciplinary treatment (IDT) — Interdisciplinary treatment (IDT)
  Arms: Interdisciplinary treatment (IDT)

SUMMARY:
This cluster randomized controlled trial evaluates whether a person-centred, AI-supported Clinical Decision Support System (CDSS) can improve outcomes and cost-effectiveness in interdisciplinary rehabilitation for people with complex chronic pain. The CDSS is designed to assist clinicians in making personalized treatment decisions within standard interdisciplinary treatment (IDT). It has been developed using machine learning models trained on real-world data from over 100,000 patients in the Swedish Quality Registry for Pain Rehabilitation (SQRP), linked to several national registers, including the National Patient Register, the Prescribed Drug Register, the Social Insurance Agency database (MiDAS), and the Cause of Death Register. This enables individualized predictions of treatment outcomes, work ability, and healthcare utilization.

The trial includes 400 adult patients with chronic pain, enrolled at 20 IDT clinics randomized to either CDSS-supported or standard IDT. The study has three phases: feasibility, effectiveness, and implementation. The primary outcome is a patient-prioritized composite single-index of health-related well-being, based on domains such as pain, sleep, physical and mental health, emotional distress, and work ability. Patients prioritize these domains together with their clinical team, enabling a person-centred assessment. Secondary outcomes include HRQoL (EQ-5D, SF-36), emotional distress (HADS), and work ability (WAI), measured at baseline, post-treatment, 6- and 12-month follow-up.

A parallel mixed-methods process evaluation will examine implementation outcomes such as usability, clinician adherence, and workflow integration, using logs, surveys (e.g., S-NoMAD), and interviews. Normalization Process Theory guides the analysis. Cost-utility will be assessed using QALYs and ICERs from a societal perspective, with long-term projections using simulation models. Results will be reported in peer-reviewed publications.

DETAILED DESCRIPTION:
This project consists of three integrated phases aimed at evaluating a machine learning-based Clinical Decision Support System (CDSS) to improve interdisciplinary rehabilitation for individuals with complex chronic pain. The evaluation encompasses feasibility, clinical effectiveness, cost-utility, and implementation in routine care. The results will be reported in multiple peer-reviewed scientific publications.

Phase 1: Development, validation, and feasibility By the end of 2025, the CDSS-developed in an ongoing project-will be ready for clinical testing. It is based on predictive models trained on registry-linked data from over 100,000 patients in the Swedish Quality Registry for Pain Rehabilitation (SQRP), linked to several national registers, including the National Patient Register, the Prescribed Drug Register, the Social Insurance Agency database (MiDAS), and the Cause of Death Register. The system provides personalized forecasts for treatment outcomes, long-term work ability, and healthcare use. A pilot cluster-RCT will be conducted at 10 clinics (5 patients per site) to evaluate feasibility outcomes such as recruitment, retention, usability, data completeness, and workflow fit. These will be assessed using structured surveys, usage data, and interviews. Outcome measures will be collected at baseline, immediately after the intervention (i.e., up to 18 weeks after baseline), and at 12-month follow-up. While a typical interdisciplinary rehabilitation program lasts 6-8 weeks, some clinics may extend the intervention up to 18 weeks (with less treatment occasions per week) due to their ordinary and existing treatment procedures at that specific clinic. Published results indicate however no significant differences in treatment outcomes based on such extended program duration (Tseli et al., 2020). No major changes to the CDSS algorithm or interface are planned during the trial.

Phase 2: Clinical effectiveness and health economic evaluation The full evaluation will be conducted through a non-registry-based cluster randomized controlled trial involving 400 patients across 20 interdisciplinary rehabilitation clinics. Outcomes will be analyzed using linear mixed-effects models adjusted for time, group, clustering, and covariates. The primary endpoint is at 12-month follow-up. Secondary outcomes will be assessed at baseline, up to 18 weeks after baseline (i.e., immediately post intervention), and at 6- and 12-month follow-up. Health economic analyses will include within-trial cost-utility evaluation (QALYs from EQ-5D and SF-36) and longer-term modelling using Markov or microsimulation methods. Both direct (healthcare) and indirect (productivity loss) costs will be included. Sensitivity analyses will address uncertainty and robustness.

Phase 3: Implementation research A mixed-methods process evaluation will examine real-world adoption, scalability, and sustainability. Data will include system logs (e.g., reach, fidelity), survey responses (S-NoMAD), and interviews with clinicians and decision-makers. Analysis is guided by Normalization Process Theory, focusing on coherence (understanding), cognitive participation (engagement), collective action (integration), and reflexive monitoring (clinical utility). This structure enables a rigorous, practice-oriented evaluation of AI support in pain rehabilitation, integrating clinical, economic, and implementation perspectives to guide responsible and scalable integration into healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 67 years
* Diagnosed with chronic non-malignant pain persisting longer than 3 months
* Pain condition includes, but is not limited to: fibromyalgia, widespread pain, back pain, neck pain, or shoulder pain
* Eligible for and referred to interdisciplinary rehabilitation (IDT) at a participating clinic
* Willing and able to participate in digital assessment and follow-up procedures
* Able to communicate and complete study materials in Swedish
* Provides written informed consent

Exclusion Criteria

* Pain caused by malignancy or cancer-related treatment
* Pain caused by systemic diseases such as rheumatoid arthritis, lupus, or other autoimmune or inflammatory conditions
* Severe psychiatric conditions interfering with study participation (e.g., untreated psychosis or severe depression requiring immediate psychiatric care)
* Documented cognitive impairment limiting ability to understand study participation or complete self-reported measures
* Currently enrolled in another interventional clinical trial that may confound the outcomes of this study
* Not expected to remain in the clinic's follow-up system for the duration of the study

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Patient-Prioritized Health-Related Well-being Composite at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  A person-centred composite score based on eight validated domains: pain intensity (NRS; 0-10), sleep problems (ISI; 0-28), physical health (SF-36 PF; 0-100), mental health (SF-36 MH; 0-100), depression and anxiety (HADS-A/D; 0-21), work ability (WAI single item; 0-10), and pain interference (single item; 0-10). At baseline, participants prioritize these domains together with the interdisciplinary treatment (IDT) team. The Clinical Decision Support System (CDSS) stores these weights. Each domain is normalized to 0-100 and combined into a weighted composite. Higher scores indicate better health-related well-being. Although composed of several scales, the outcome is reported as a single, aggregated primary measure.

SECONDARY OUTCOMES:
Change from Baseline in Pain Intensity (NRS) at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  Measured using the Numeric Rating Scale (NRS, 0-10), where 0 = no pain and 10 = worst imaginable pain. Participants report average pain over the last seven days. A reduction in score indicates clinical improvement.
Change from Baseline in Sleep Problems Measured by the Insomnia Severity Index (ISI) at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  The ISI assesses perceived sleep difficulties through seven items. Total scores range from 0 to 28, with higher values indicating more severe insomnia. A lower score reflects improved sleep quality.
Change from Baseline in Physical Health Functioning (SF-36 PF) at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  Measured using the SF-36 Physical Functioning subscale (10 items). Scores range from 0 to 100, with higher scores representing better physical functioning.
Change from Baseline in Mental Health (SF-36 MH) at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  Measured using the SF-36 Mental Health subscale (5 items). Scores range from 0 to 100; higher values indicate better mental well-being.
Change from Baseline in Emotional Distress Measured by the Hospital Anxiety and Depression Scale (HADS) at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  The HADS includes two 7-item subscales for anxiety and depression. Each subscale ranges from 0 to 21; higher scores indicate greater emotional distress.
Change from Baseline in Work Ability Measured by the Work Ability Index (WAI) Single Item at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  Assessed via the single-item WAI: "Current work ability compared to lifetime best", scored from 0 (completely unable to work) to 10 (work ability at its best).
Change from Baseline in Pain Interference in Daily Life at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  Measured using validated items adapted from the Multidimensional Pain Inventory or equivalent, reflecting the extent to which pain disrupts everyday activities. Scores are standardized from 0 (no interference) to 100 (maximum interference).
Change from Baseline in Physical Activity Measured by the Exercise Vital Sign (EVS) at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  The EVS includes two questions: (1) days per week of moderate-to-strenuous activity, and (2) average minutes per day. The product gives total minutes/week. Validated against objective activity measures.
Treatment Expectations at Baseline | At enrollment (baseline) only.
  A single-item self-report question regarding the individual's expectation of treatment benefit, rated on a Likert scale from "no improvement expected" to "complete recovery expected".
Change from Baseline in Sick Leave Status at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  Self-reported current sick leave status (full-time, part-time, or not on leave). Changes over time reflect return-to-work or ongoing sick leave status.
Change from Baseline in Self-Reported Medication Use at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  Captured through a validated web-based tool. Participants report medication name (text), dose (mg), frequency (time/day), and form (e.g. tablet). Variables are analyzed separately using descriptive statistics and longitudinal methods to assess changes in medication use over time.
Change in Cost-Utility at 24 Months (EQ-5D-5L) | (1) Up to 18 weeks after baseline, (2) 12 months, and (3) 24 months after treatment completion.
  Measured in Quality-Adjusted Life Years (QALYs) derived from the EuroQol 5-Dimension 5-Level (EQ-5D-5L) instrument using standard value sets. The Incremental Cost-Effectiveness Ratio (ICER) will be calculated as the ratio of the difference in costs to the difference in health outcomes (QALYs gained), comparing the intervention to the control. ICER provides a summary measure of the additional cost required to gain one additional unit of health benefit.
  EQ-5D index scores typically range from below zero (e.g., -0.594 in the UK value set) to 1.000, or from 0.296 to 1.000 using the Swedish experience-based value set, where higher values indicate better health-related quality of life.
Change in Cost-Utility at 24 Months (RAND SF-36) | (1) Up to 18 weeks after baseline, (2) 12 months, and (3) 24 months after treatment completion.
  Measured using the RAND 36-Item Health Survey (RAND SF-36), which assesses physical and mental health across eight domains. Each domain score ranges from 0 to 100, with higher scores indicating better health status. A cost-utility analysis will also be performed using utility estimates derived from RAND SF-36, and an ICER will be calculated accordingly. ICER will be interpreted as the additional cost per unit of utility gained, based on mapped utility values. (Note: Mapping algorithms may be applied to derive utility weights from RAND SF-36, subject to validation.)

OTHER OUTCOMES:
Change in Sickness Absence (Register-Based) at 12 Months | From 5 years before baseline to 5 years after the 12-month follow-up.
  Data obtained from the Swedish Social Insurance Agency (MiDAS) detailing sickness absence (full- or part-time) in number of net days. Fewer days indicate clinical or occupational improvement. Scores range from 0 to an open upper limit, where 0 indicates no sickness absence and higher values indicate more days of absence.
Change in Total Prescribed Medication Volume (Register-Based) at 12 Months | From 5 years before baseline to 5 years after the 12-month follow-up.
  Data will be extracted from the Swedish Prescribed Drug Register. Medication volume will be calculated using the Defined Daily Dose (DDD) methodology, as defined by the World Health Organization (WHO). For each prescribed medication, the total number of dispensed units will be converted into DDDs based on the standard daily maintenance dose for its main indication in adults. The total DDDs per individual will be summed across all medications to reflect overall pharmacological treatment intensity. Scores range from 0 to no predefined upper limit, where higher values indicate greater medication burden.
Change in Comorbidity Burden Over Time | From 5 years before baseline to 5 years after the 12-month follow-up.
  Comorbidity burden will be derived from the Swedish National Patient Register using established ICD-10 codes. A validated multimorbidity index (e.g., the Charlson Comorbidity Index or a count of chronic conditions) will be calculated for each individual at multiple time points. Higher scores reflect a greater burden of comorbid disease. Scores typically range from 0 (no comorbid conditions) to 15 or more, depending on the index used and the number/severity of conditions present.
Change in Pain Location Complexity Over Time | From 5 years before baseline to 5 years after the 12-month follow-up.
  Self-reported pain drawings will be analyzed to determine the number of distinct anatomical pain locations reported by each participant. This measure reflects the spatial complexity of pain presentation. Scores range from 0 (no reported pain) to approximately 36, based on a standardized body map divided into predefined regions. Higher scores indicate more widespread or complex pain distribution.
Change from Baseline in Pain Acceptance as Measured by the Chronic Pain Acceptance Questionnaire (CPAQ-8) at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  CPAQ-8 includes 8 items (score 0-6 per item), total score 0-48. Higher scores represent greater acceptance of pain.
Change from Baseline in Fear-Avoidance Beliefs as Measured by the Tampa Scale of Kinesiophobia (TSK) at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  TSK (13 items) total score range: 13-52. Higher scores indicate greater fear of movement. Decreases reflect improvement in pain-related fear.
Change from Baseline in Pain Catastrophizing at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  Measured using the Pain Catastrophizing Scale (PCS). Scores range from 0 to 52; higher scores denote greater catastrophizing.
Change from Baseline in Pain Self-Efficacy at 12 Months | (1) Baseline, (2) up to 18 weeks after baseline*, and (3) 12-month follow-up. (*Most programs last 6-8 weeks, but some clinics extend to 18 weeks (fewer sessions/week) due to existing routine practice).
  Assessed using the Pain Self-Efficacy Questionnaire (PSEQ), score range 0-60. Higher scores reflect greater confidence in functioning despite pain.

CONTACTS AND LOCATIONS:
Overall Officials: Björn O Äng, Professor, Principal Investigator — Dalarna University
Locations (1):
- Dalarna University, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) may be shared upon reasonable request, pending legal and ethical approval. The research team is currently reviewing the feasibility of data sharing under Swedish regulations (e.g., GDPR).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data (IPD) and supporting documentation will be made available beginning 12 months after publication of the primary results. Access will be granted upon reasonable request and subject to approval by the principal investigator and relevant ethical and legal review, in accordance with Swedish data protection regulations (e.g., GDPR).
Access Criteria: Access to de-identified individual participant data (IPD) and supporting documentation may be granted to qualified researchers affiliated with academic or healthcare institutions, for ethically approved research purposes. Requests must include a detailed research proposal and ethical approval from an appropriate Swedish or EU-recognized ethics review board. All requests will be reviewed by the principal investigator and the responsible data controller at the host institution. A data sharing agreement must be signed. Data access will be provided through secure transfer mechanisms, in full compliance with the Swedish Patient Data Act (PDL) and the General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Elf M, Nordmark S, Lyhagen J, Lindberg I, Finch T, Aberg AC. The Swedish version of the Normalization Process Theory Measure S-NoMAD: translation, adaptation, and pilot testing. Implement Sci. 2018 Dec 4;13(1):146. doi: 10.1186/s13012-018-0835-5. PMID 30509289
- [Background] Edwards RR, Schreiber KL, Dworkin RH, Turk DC, Baron R, Freeman R, Jensen TS, Latremoliere A, Markman JD, Rice ASC, Rowbotham M, Staud R, Tate S, Woolf CJ, Andrews NA, Carr DB, Colloca L, Cosma-Roman D, Cowan P, Diatchenko L, Farrar J, Gewandter JS, Gilron I, Kerns RD, Marchand S, Niebler G, Patel KV, Simon LS, Tockarshewsky T, Vanhove GF, Vardeh D, Walco GA, Wasan AD, Wesselmann U. Optimizing and Accelerating the Development of Precision Pain Treatments for Chronic Pain: IMMPACT Review and Recommendations. J Pain. 2023 Feb;24(2):204-225. doi: 10.1016/j.jpain.2022.08.010. Epub 2022 Oct 2. PMID 36198371
- [Background] May CR, Mair F, Finch T, MacFarlane A, Dowrick C, Treweek S, Rapley T, Ballini L, Ong BN, Rogers A, Murray E, Elwyn G, Legare F, Gunn J, Montori VM. Development of a theory of implementation and integration: Normalization Process Theory. Implement Sci. 2009 May 21;4:29. doi: 10.1186/1748-5908-4-29. PMID 19460163
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Gronkvist R, Vixner L, Ang B, Grimby-Ekman A. Measurement Error, Minimal Detectable Change, and Minimal Clinically Important Difference of the Short Form-36 Health Survey, Hospital Anxiety and Depression Scale, and Pain Numeric Rating Scale in Patients With Chronic Pain. J Pain. 2024 Sep;25(9):104559. doi: 10.1016/j.jpain.2024.104559. Epub 2024 May 10. PMID 38734041
- [Background] Sjoberg V, Westergren J, Monnier A, Lo Martire R, Hagstromer M, Ang BO, Vixner L. Wrist-Worn Activity Trackers in Laboratory and Free-Living Settings for Patients With Chronic Pain: Criterion Validity Study. JMIR Mhealth Uhealth. 2021 Jan 12;9(1):e24806. doi: 10.2196/24806. PMID 33433391
- [Background] Sjoberg V, Monnier A, Tseli E, LoMartire R, Hagstromer M, Bjork M, Ang B, Vixner L. Feasibility and acceptability of design and conduct of a registry-based randomised clinical trial evaluating eVIS as a digital support for physical activity in interdisciplinary pain rehabilitation programs: A randomised pilot study. Digit Health. 2024 Nov 25;10:20552076241299648. doi: 10.1177/20552076241299648. eCollection 2024 Jan-Dec. PMID 39600393
- [Background] Westergren J, Sjoberg V, Vixner L, Nyberg RG, Moulaee Conradsson D, Monnier A, LoMartire R, Enthoven P, Ang BO. Acute exercise as active inference in chronic musculoskeletal pain, effects on gait kinematics and muscular activity in patients and healthy participants: a study protocol for a randomised controlled laboratory trial. BMJ Open. 2023 May 31;13(5):e069747. doi: 10.1136/bmjopen-2022-069747. PMID 37258077
- [Background] LoMartire R, Ang BO, Gerdle B, Vixner L. Psychometric properties of Short Form-36 Health Survey, EuroQol 5-dimensions, and Hospital Anxiety and Depression Scale in patients with chronic pain. Pain. 2020 Jan;161(1):83-95. doi: 10.1097/j.pain.0000000000001700. PMID 31568237
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Strom P, Kartasalo K, Olsson H, Solorzano L, Delahunt B, Berney DM, Bostwick DG, Evans AJ, Grignon DJ, Humphrey PA, Iczkowski KA, Kench JG, Kristiansen G, van der Kwast TH, Leite KRM, McKenney JK, Oxley J, Pan CC, Samaratunga H, Srigley JR, Takahashi H, Tsuzuki T, Varma M, Zhou M, Lindberg J, Lindskog C, Ruusuvuori P, Wahlby C, Gronberg H, Rantalainen M, Egevad L, Eklund M. Artificial intelligence for diagnosis and grading of prostate cancer in biopsies: a population-based, diagnostic study. Lancet Oncol. 2020 Feb;21(2):222-232. doi: 10.1016/S1470-2045(19)30738-7. Epub 2020 Jan 8. PMID 31926806
- [Background] Moazemi S, Vahdati S, Li J, Kalkhoff S, Castano LJV, Dewitz B, Bibo R, Sabouniaghdam P, Tootooni MS, Bundschuh RA, Lichtenberg A, Aubin H, Schmid F. Artificial intelligence for clinical decision support for monitoring patients in cardiovascular ICUs: A systematic review. Front Med (Lausanne). 2023 Mar 31;10:1109411. doi: 10.3389/fmed.2023.1109411. eCollection 2023. PMID 37064042
- [Background] Granviken F, Vasseljen O, Bach K, Jaiswal A, Meisingset I. Decision Support for Managing Common Musculoskeletal Pain Disorders: Development of a Case-Based Reasoning Application. JMIR Form Res. 2024 May 10;8:e44805. doi: 10.2196/44805. PMID 38728686
- [Background] Tseli E, LoMartire R, Vixner L, Grooten WJA, Gerdle B, Ang BO. What Is the Effectiveness of Different Duration Interdisciplinary Treatment Programs in Patients with Chronic Pain? A Large-Scale Longitudinal Register Study. J Clin Med. 2020 Aug 29;9(9):2788. doi: 10.3390/jcm9092788. PMID 32872448
- [Background] Gerdle B, Akerblom S, Brodda Jansen G, Enthoven P, Ernberg M, Dong HJ, Stalnacke BM, Ang BO, Boersma K. Who benefits from multimodal rehabilitation - an exploration of pain, psychological distress, and life impacts in over 35,000 chronic pain patients identified in the Swedish Quality Registry for Pain Rehabilitation. J Pain Res. 2019 Mar 7;12:891-908. doi: 10.2147/JPR.S190003. eCollection 2019. PMID 30881099
- [Background] LoMartire R, Bjork M, Dahlstrom O, Constan L, Frumento P, Vixner L, Gerdle B, Ang BO. The value of interdisciplinary treatment for sickness absence in chronic pain: A nationwide register-based cohort study. Eur J Pain. 2021 Nov;25(10):2190-2201. doi: 10.1002/ejp.1832. Epub 2021 Jul 20. PMID 34189810
- [Background] Dragioti E, Evangelou E, Larsson B, Gerdle B. Effectiveness of multidisciplinary programmes for clinical pain conditions: An umbrella review. J Rehabil Med. 2018 Sep 28;50(9):779-791. doi: 10.2340/16501977-2377. PMID 30132012
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain: Cochrane systematic review and meta-analysis. BMJ. 2015 Feb 18;350:h444. doi: 10.1136/bmj.h444. PMID 25694111
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143
- [Background] Gatchel RJ, McGeary DD, McGeary CA, Lippe B. Interdisciplinary chronic pain management: past, present, and future. Am Psychol. 2014 Feb-Mar;69(2):119-30. doi: 10.1037/a0035514. PMID 24547798
- [Background] Leadley RM, Armstrong N, Lee YC, Allen A, Kleijnen J. Chronic diseases in the European Union: the prevalence and health cost implications of chronic pain. J Pain Palliat Care Pharmacother. 2012 Dec;26(4):310-25. doi: 10.3109/15360288.2012.736933. PMID 23216170
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. Chronic pain as a symptom or a disease: the IASP Classification of Chronic Pain for the International Classification of Diseases (ICD-11). Pain. 2019 Jan;160(1):19-27. doi: 10.1097/j.pain.0000000000001384. PMID 30586067
- [Background] Kaiser U, Treede RD, Sabatowski R. Multimodal pain therapy in chronic noncancer pain-gold standard or need for further clarification? Pain. 2017 Oct;158(10):1853-1859. doi: 10.1097/j.pain.0000000000000902. No abstract available. PMID 28328572
- [Background] Wiens J, Shenoy ES. Machine Learning for Healthcare: On the Verge of a Major Shift in Healthcare Epidemiology. Clin Infect Dis. 2018 Jan 6;66(1):149-153. doi: 10.1093/cid/cix731. PMID 29020316
- [Background] Goldstein P, Ashar Y, Tesarz J, Kazgan M, Cetin B, Wager TD. Emerging Clinical Technology: Application of Machine Learning to Chronic Pain Assessments Based on Emotional Body Maps. Neurotherapeutics. 2020 Jul;17(3):774-783. doi: 10.1007/s13311-020-00886-7. PMID 32767227
- [Background] Edwards RR, Dworkin RH, Turk DC, Angst MS, Dionne R, Freeman R, Hansson P, Haroutounian S, Arendt-Nielsen L, Attal N, Baron R, Brell J, Bujanover S, Burke LB, Carr D, Chappell AS, Cowan P, Etropolski M, Fillingim RB, Gewandter JS, Katz NP, Kopecky EA, Markman JD, Nomikos G, Porter L, Rappaport BA, Rice ASC, Scavone JM, Scholz J, Simon LS, Smith SM, Tobias J, Tockarshewsky T, Veasley C, Versavel M, Wasan AD, Wen W, Yarnitsky D. Patient phenotyping in clinical trials of chronic pain treatments: IMMPACT recommendations. Pain. 2016 Sep;157(9):1851-1871. doi: 10.1097/j.pain.0000000000000602. PMID 27152687
- [Background] Whitehead SJ, Ali S. Health outcomes in economic evaluation: the QALY and utilities. Br Med Bull. 2010;96:5-21. doi: 10.1093/bmb/ldq033. Epub 2010 Oct 29. PMID 21037243
- [Background] James S, Rao SV, Granger CB. Registry-based randomized clinical trials--a new clinical trial paradigm. Nat Rev Cardiol. 2015 May;12(5):312-6. doi: 10.1038/nrcardio.2015.33. Epub 2015 Mar 17. PMID 25781411
- [Background] Maramba I, Chatterjee A, Newman C. Methods of usability testing in the development of eHealth applications: A scoping review. Int J Med Inform. 2019 Jun;126:95-104. doi: 10.1016/j.ijmedinf.2019.03.018. Epub 2019 Mar 31. PMID 31029270
- [Background] IASP, Task Force on Multimodal Pain Treatment Defines Terms for Chronic Pain Care. 2017.
- [Background] SBU, Multimodal rehabilitering vid långvarig ländryggssmärta. 2015: Stockholm.
- [Background] SBU, Multimodala och interdisciplinära behandlingar vid långvarig smärta: en systematisk översikt och utvärdering av effekter på hälsa och hälsoekonomiska aspekter. 2021: Stockholm.
- [Background] SBU, Behandling och rehabilitering vid fibromyalgi: en systematisk översikt och utvärdering av effekter på hälsa., 2021: Stockholm.
- [Background] Hopp, W.J., et al., Big Data and the Precision Medicine Revolution. Prod Oper Manag, 2018. 27(9).
- [Background] Ware, J.E., et al., SF-36 health survey: manual and interpretation guide 1993, Quality Metric.
- [Background] Swedish Social Insurance Agency, Proposal of outcome measures of return to work. Rep. 2016:9
- [Background] Dey, A., Machine Learning Algorithms : A Review. IJCSIT, 2016. 7(3): p. 1174.
- See also: Research project/group — https://www.du.se/en/research/research-project/?projectid=110